CLINICAL TRIAL: NCT03835091
Title: Use of BRASS in Sedated Critically-ill Patients as a Predictable Mortality Factor
Acronym: BRASS-ICU
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18167
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Brainstem Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with mechanical ventilation and sedation: All patient hospitalized in intensive care under sedation and mechanical ventilation without neurologic disorder
  Interventions: Other: BRASS score

INTERVENTIONS:
Other: BRASS score — Brainstem response on neurologic examination

SUMMARY:
Sedation is used for 30 to 70 % of all intensive care unit (ICU) patients. Deep sedation can be used for lot of disease like acute respiratory distress syndrome, septic shock.

Deep sedation was defined by RASS (Richmond Assessment Sedation Scale) below -3.

Deep sedation can be associated with increased mortality, length stay, duration of mechanical ventilation, acute brain dysfunction.

The french exploration neurologic group in ICU developed a score used Brainstem response patterns in patient deeply sedated by midazolam and showed that a high BRASS score is associated with high mortality at day 28.

The investigators think that BRASS score isn't associated with the medication used for sedation.

In this study the investigators included all patients sedated independently of medication used for sedation, we also excluded patient with neurologic disorder.

The main objective is to shown that high BRASS score at admission of patient without neurologic disorder sedated is predictive of 28-day mortality.

DETAILED DESCRIPTION:
Sedation is used for 30 to 70 % of all intensive care unit (ICU) patients. Deep sedation can be used for lot of disease like acute respiratory distress syndrome, septic shock.

Deep sedation was defined by RASS (Richmond Assessment Sedation Scale) below -3.

Deep sedation can be associated with increased mortality, length stay, duration of mechanical ventilation, acute brain dysfunction.

The french exploration neurologic group in ICU developed a score used Brainstem response patterns in patient deeply sedated by midazolam and showed that a high BRASS score is associated with high mortality at day 28.

The investigators think that BRASS score isn't associated with the medication used for sedation.

In this study the investigators included all patients sedated independently of medication used for sedation, we also excluded patient with neurologic disorder.

The main objective is to shown that high BRASS score at admission of patient without neurologic disorder sedated is predictive of 28-day mortality.

The BRASS score will be done in the 6 hours within admission. The Richmond Assessment Sedation Scale (RASS) and Full Outline of unresponsiveness (FOUR) will be performed.

The patient characteristic's will be recorded (sex, age, Simplified Acute Physiology Score II (SAPS II), medical or surgical admission, diagnosis at ICU admission (ARDS, sepsis,…), the reason of initiation of mechanical ventilation, the reason of sedation (agitation, analgesia, asynchrony with ventilator).

The medication for sedation and the level at time of examination, the time between admission and examination will be recorded.

For the outcome, the duration of mechanical ventilation, the duration of sedation administration, the occurrence of delirium evaluated by Confusion Assessment Method- intensive care unit (CAM-ICU), the length stay in ICU, death at day 28 and 90 will be reported.

ELIGIBILITY:
Inclusion Criteria:

Patient more than 18 years Hospitalized in ICU Without neurologic disorder and/or neurologic pattern Under sedation and mechanical ventilation

Exclusion Criteria:

Patients with legal protection No affiliation with the French Health Care system Ongoing pregnancy Inability to obtain consent Not to resuscitate decision Neurologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be included in this study are patients with sedation and on mechanical ventilation, without neurologic disorder
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
mortality within 28 days after ICU admission | 28 days
  percentage of patients who died within 28 days after admission

SECONDARY OUTCOMES:
mortality within 90 days after ICU admission | 90 days
  percentage of patients who died within 90 days after admission
ICU Stay | 6 months
  mean of duration of ICU stay
Delirium | 6 months
  percentage of patients with delirium
duration on mechanical ventilation | 6 months
  mean of duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Derived] Legros V, Mourvillier B, Floch T, Candelier Q, Rosman J, Lafont B, Farkas JC, Bard M, Kanagaratnam L, Mateu P. Use of BRASS in sedated critically-ill patients as a predictable mortality factor: BRASS-ICU. Neurol Res. 2021 Apr;43(4):283-290. doi: 10.1080/01616412.2020.1849901. Epub 2020 Nov 19. PMID 33208055